CLINICAL TRIAL: NCT03064256
Title: EFFECT OF AEROBIC PHYSICAL TRAINING WITH DETERMINED INTENSITY FOR THE PROTOCOL OF DOUBLE EXHAUSTIVE EFFORTS IN THE AUTONOMICAL MODULATION OF THE HEART FREQUENCY OF PATIENTS WITH SYSTEMIC ARTERIAL HYPERTENSION
Brief Title: Aerobic Physical Training and Heart Rate Variability in Hypertersion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Campinas, Brazil (Other)
Collaborators: Medical Outpatient Vlinic of the Government of the State of São Paulo (Unknown)
Responsible Party: Principal Investigator, Taís Mendes de Camargo, PhD student, University of Campinas, Brazil
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 865.096
Record Dates: First submitted 2017-02-19; First posted 2017-02-27 (Actual); Last update posted 2017-02-27 (Actual); Status verified 2017-02

CONDITIONS: Autonomic Nervous System Diseases
Keywords: Exercisy therapy; Hypertension; Physiopathology; Heart rate; Nonlinear dynamics
MeSH Terms: conditions — Autonomic Nervous System Diseases; Hypertension

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Physical training program (Experimental): Intervention participants are submitted to supervised aerobic physical training at the predetermined intensity, which is composed of three weekly sessions, lasting one hour, over a period of 12 weeks.
  All sessions were started with stretches for lower and upper limbs lasting 10 minutes for warm-up, and after trekking on treadmill using the predetermined critical velocity (Vcrit). The exercises were completed with cooling of the muscle groups for one minute still on the treadmill, plus 10 minutes of relaxation exercises on the mat at the end of aerobic exercise.
  Interventions: Behavioral: Physical training program
- Control Group (No Intervention): Control participants receive routine outpatient care for a 12-week period.

INTERVENTIONS:
Behavioral: Physical training program — Physical training program consisted of three weekly sessions lasting up to one hour over a period of twelve weeks. and will be carried out respecting the traditional training principles: biological individuality, Specificity, overload, adaptation and reversibility
  Arms: Physical training program
Behavioral: Physical training program — All sessions were started with stretches for lower and upper limbs lasting 10 minutes for warm-up, and after trekking on treadmill using the predetermined critical velocity (Vcrit). The exercises were completed with cooling of the muscle groups for one minute still on the treadmill, plus 10 minutes of relaxation exercises on the mat at the end of aerobic exercise.
  Arms: Physical training program

SUMMARY:
This study compared the changes in the cardiovascular, hemodynamic and metabolic variables of hypertensive patients who received aerobic physical training with intensity determined by the protocol of double non-exhaustive efforts (DENE) with that of patients who received routine outpatient care 12 weeks after Entry into the study. 63 men and women participated in the study and were allocated in the intervention group (n = 42) and control group (n = 21).The following were performed: Cardiopulmonary exercise test (TECP) for evaluation of peak oxygen consumption (VO2peak), oxygen pulse and double product; DENE protocol for the determination of the intensity of the training. It was obtained the recording of the intervals between consecutive heart beats (iRR) to evaluate the autonomic modulation of the heart rate. Body mass index, waist circumference (AC), hip circumference (CQ) and Waist / hip ratio (WHR) were measured.

DETAILED DESCRIPTION:
The study was designed to compare changes in the cardiovascular, hemodynamic and metabolic variables of hypertensive patients who received aerobic physical training with intensity determined by the DENE protocol with that of patients who received routine ambulatory care 12 weeks after entering the study.

Sixty-three hypertensive men and women, divided into the intervention group (GI) (n=42) and the control group (n = 21) participated in the study.

All procedures were performed by trained researchers and qualified staff and the evaluations and intervention were performed at the specialty medical outpatient clinic.

After agreeing to participate in the study, we collected sociodemographic and clinical data, body mass index (BMI), waist circumference (WC) and waist / hip ratio (WHR). The participants were submitted to the cardiopulmonary exercise test (TECP), to evaluate the peak oxygen consumption (VO2peak), oxygen pulse and double product. Between one and seven days after TECP, consecutive heart rate intervals (iRR) were recorded for evaluation of autonomic heart rate modulation using a Polar model RS800CX (Polar Electro Co.Ltda Kempele, Finland). . The DENE protocol for determining the intensity of the training was applied in the GI to determine the training intensity in the treadmill. Intervention participants underwent supervised aerobic physical training at the pre-determined intensity, which consisted of three weekly sessions, lasting one hour, over a period of 12 weeks. Control participants receive routine care from the outpatient clinic for the same period. At the end of the 12 weeks, measures, recording of the iRR intervals, oxygen pulse, double product, BMI, waist circumference (AC), hip circumference (QC) and waist / hip ratio (WHR) were obtained. All subjects were previously informed about the procedures Signed a free and informed consent form. The project was approved by the Commission of Research Committee of the Institution with the number 086.096 / 14.

ELIGIBILITY:
Inclusion Criteria:

* SBP ≤ 180 mmHg and DBP ≤ 110 mmHg)
* low risk for physical training.

Exclusion Criteria:

* obesity III
* musculoskeletal conditions
* peripheral neuropathy
* Parkinson's disease.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2014-11-14 (Actual); Primary Completion 2015-12-21 (Actual); Study Completion 2017-01-16 (Actual)

PRIMARY OUTCOMES:
Heart rate variability will be measured by nonlinear methods in hypertensive patients to observe changes in baseline values after 12 weeks. | Finalized study (12 weeks)
  A heart rate meter RS800CX (Polar Electro Co.Ltda. Kempele, Finland) is used to obtain HR and R-R (iR-R) intervals. The iR-Rs are captured from a tape with a coded transmitter placed in the chest region at the 5th intercostal space and transmitted to the cardiofrequency meter where they are recorded

SECONDARY OUTCOMES:
The peak oxygen consumption (mL / kg · min) will be measured by ergospirometry in hypertensive patients to observe changes in baseline values after 12 weeks. | Finalized study (12 weeks)
  Cardiopulmonary exercise test used to determine peak oxygen consumption to exercise .
The double product (mmHg) will be measured by ergospirometry in hypertensive patients to observe changes in baseline values after 12 weeks. | Finalized study (12 weeks)
  Cardiopulmonary exercise test used to determine double produc to exercise .
The oxigen pulse (ml/heart rate) will be measured by ergospirometry in hypertensive patients to observe changes in baseline values after 12 weeks. | Finalized study (12 weeks)
  Cardiopulmonary exercise test used to determine oxigen pulse to exercise .